CLINICAL TRIAL: NCT04983017
Title: Randomized, Double-Blinded, Placebo-Controlled Study With Immunotype Specific Dietary Supplements to Improve Inflammatory Age® by Edifice Health
Brief Title: 2021 PMT iAge® Intervention Trial by Edifice Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was no significant difference between placebo and control.
Sponsor: Edifice Health (Industry)
Responsible Party: Principal Investigator, Lizellen La Follette, MD, OBGYN, Edifice Health
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: EH_21_01_PMT_iAge_INT
Record Dates: First submitted 2021-07-26; First posted 2021-07-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Inflammation; Inflammaging
Keywords: inflammatory age (iAge®); immunosenescence; immune phenotyping; systemic chronic inflammation
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Participants will receive a formulation of dietary supplements based on the iAge test. Different formulations contain different combinations of dietary supplements.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplements (Active Comparator): Dietary supplements are either (1) designated as Generally Recognized As Safe (GRAS) by the Food and Drug Administration or (2) compounds at similar concentrations to those found in foods.
  Interventions: Dietary Supplement: Dietary supplement
- Placebo (Placebo Comparator): Placebo-matched formulations
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary supplement — iron bisglycinate manganese chloride vitamin D2 guar gum indole-3-carbinol L-methionine piceatannol biotin caffeine beta-carotene lutein zinc sulfate
  Arms: Dietary supplements
Other: Placebo — Matched Placebo to Intervention
  Arms: Placebo

SUMMARY:
This is a decentralized, double-blind, randomized, placebo-controlled study to assess the effectiveness of different dietary supplements in decreasing systemic chronic inflammation (SCI) and lowering inflammatory age (iAge®). iAge® is a metric for age-related chronic inflammation and immune function decline calculated from a standard blood draw utilizing immune phenotyping and artificial intelligence algorithms. SCI is a natural process that occurs within the body. It is believed to accelerate the process of biological aging. As opposed to acute inflammation, iAge® is not a reflection of illness, infection, trauma or injury. It naturally occurs in the ambulatory healthy population as we age as a function of the body.

This study will use immunotype specific dietary supplement formulations to improve a participant's Inflammatory Age® (iAge®).

DETAILED DESCRIPTION:
This decentralized, double-blind, randomized, placebo-controlled study will identify interventions that may lower a participant's inflammatory age (iAge®) and will increase the number of participants with objective and subjective health information that have associated iAge® scores. The study will also (1) correlate secondary endpoints with baseline and subsequent iAge® scores, (2) confirm the compatibility of the iAge® test with the Tasso device, ADX100 or ViveBio home blood collection systems, and (3) confirm the compatibility of the iAge® test with saliva home sample collection kit.

Ambulatory adults, 18 years old and over of diverse ethnicities will be invited to participate in this study from a single site in Marin County. We will choose an equal number of male and female participants by selecting households within a 60 mile radius of the study site.

The study involves fasting blood sample collection to measure and characterize immunomes and inflammatory biomarkers, metabolites, lipid panel, hemoglobin, hemoglobin A1C, and high-sensitivity c-reactive protein (hsCRP). Participants will be asked to provide a blood sample by routine venipuncture at Baseline and approximately 2, 4 and 7 months after the start of the dietary supplement/placebo.

Participants will be given interventions to be taken daily based on their associated immunogroup cluster after each iAge® test is completed. Participants can continue on their current supplements but should not start any new supplements except those given by the study. This study has a different intervention for nine of the ten immunotype clusters. All interventions are i) generally recognized as safe (GRAS) or ii) from compounds at similar concentrations to those found in foods. Participants will be placed in one of ten immunotype clusters after each iAge® test and randomized either to a placebo or the given formulation to be taken once daily (either one, two or three pills depending on the formulation). A participant who changes his/her immunotype cluster after a follow up iAge® test will be given a new dietary intervention (or placebo based on their previous category).

All participants will also be given a Whoop wearable watch to collect information on strain, sleep and heart rate variability. Participants will be asked to complete questionnaires assessing mood, stress level, well-being, cognition, health and lifestyle. We will also obtain the following measurements: (1) Height and weight, (2) blood pressure, (3) waist and hip measurements, (4) pulse wave velocity (PWV) to measure arterial stiffness (5) timed up and go to assess frailty and (6) facial and scalp photos.

A gut microbiome sampling using a third party kit for fecal collection will be obtained at each designated time point from those participants who agree to have fecal sample collection. A subset of participants will have the following procedures done at any time point during the study: (1) saliva collection, (2) heel bone density, (3) audiometry test, (4) home blood sample collection using the Tasso device, ADX100, and ViveBio device.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Ambulatory
* Willing and able to comply with the study protocol

Exclusion Criteria:

* Participants with any condition that may preclude venipuncture or venous blood draws will be excluded.
* Participants with known allergies to interventions will be removed from the study.
* Vulnerable subjects including children, employees and those with cognitive disabilities will not be included in this study.
* Male participants on iron supplementation
* Participants on >1 mg manganese, >5 mg biotin
* Pregnant women
* Nursing women
* Membership in the clinical study team
* Any condition that might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol

At the time of enrollment:

* Active systemic or serious concurrent illness
* History of immunodeficiency
* Any known or suspected impairment of immunologic function
* Diabetes mellitus treated with any diabetic medication
* Moderate to severe renal disease
* Blood pressure greater than 140/90
* Chronic hepatitis B or C
* Recent or current use of immunosuppressive medication
* Malignancy other than squamous cell or basal cell skin cancer, including solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia, which might jeopardize volunteer safety or compliance with the protocol
* Autoimmune disease
* Auto-inflammatory disease
* History of blood dycrasias or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
* Use of any anticoagulation medication
* A medical or psychiatric condition or occupational responsibilities that would preclude subject compliance with the protocol
* History of Guillain-Barre syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory age (iAge®) scores from Baseline to end of study intervention | Measured at Baseline, Day 50, Day 120 and Day 210
  Measurement of iAge® scores in all study participants. Peripheral blood samples will be collected, processed and analyzed and iAge is measured using standardized procedures, immune phenotyping and artificial intelligence algorithms.

SECONDARY OUTCOMES:
Change in immune protein biomarkers from Baseline to end of study intervention | Measured at Baseline, Day 50, Day 120 and Day 210
  Blood sample measurements of the levels of the biomarkers Eotaxin-1 (CCL11), Interferon-gamma, Growth Regulated Oncogene-alpha, Monokine Induced by Gamma Interferon (MIG) and TNF-related Apoptosis Inducing Ligand (TRAIL)
Change in values for hemoglobin, A1C, high sensitivity C-reactive protein (hs-CRP), and lipid panel from Baseline to end of study intervention | Measured at Baseline, Day 50, Day 120 and Day 210
  Blood samples measured for hemoglobin, A1C, hs-CRP, and lipid panel
Anthropometric and metabolic measurements from Baseline to end of study intervention | Measured at Baseline, Day 50, Day 120 and Day 210
  Measurement of height, weight, body mass index (BMI), waist-to-hip ratio
Change in cardiovascular health from Baseline to end of study intervention | Measured at Baseline, Day 50, Day 120 and Day 210
  Measurement of blood pressure, pulse wave velocity using the Whithings Cardio device and heart rate variability with the Whoop wearable
Correlation of iAge score with ankle bone density score | Measured at a single time point during the duration of the study
  Measurement of ankle bone density using the GE Achilles Lunar Express ultrasonometer
Correlation of iAge score with hearing test score | Measured at a single time point during the duration of the study
  Measurement of hearing acuity using the Shoebox Audiometry System
Change in frailty and mobility from Baseline to end of study intervention | Measured at Baseline and Day 210
  Timed Up and Go (TUG) test will be use to measure the length of time in seconds it takes for the participant to stand from a chair, walk 3 meters, turn around and sit back in the chair. TUG is a simple sensitive test to assess mobility, balance, walking ability, and fall risk in older adults.

OTHER OUTCOMES:
Track fitness performance biometrics from Baseline to end of study intervention | Measured at Baseline, Day 50, Day 120 and Day 210
  Measurement and monitoring of sleep, strain, and heart rate variability using the WHOOP wearable device
Assessment of skin and scalp health from Baseline to end of study intervention | Measured at Baseline, Day 50, Day 120 and Day 210
  Facial and scalp photos will be taken using an iPAD
Saliva sample collection | Measured at Baseline in a subset of participants
  General and oral health assessment through saliva sample collection in a subset of participants
Changes in the gut microbiome at Baseline to end of study intervention in a subset of participants | Measured at a single time point during the duration of the study in a subset of participants
  Evaluate changes in the gut microbiome using the Thryve Gut Health Test Kit to collect stool samples
Correlation of standard venipuncture with at-home Tasso, ADX100m and ViveBio collection system in predicting iAge | Measured at Baseline in a subset of participants
  Capillary blood collection using the at-home Tasso, ADX100 and ViveBio collection system in a subset of study participants
Changes in metabolomic profile | Measured at Baseline, Day 50, Day 120 and Day 210 in a subset of participants
  In a subset of participants, metabolite analysis of blood plasma using high-throughput technology
Skin pH | Measured at Baseline, Day 50, Day 120 and Day 210 in a subset of participants
  Skin pH probe

CONTACTS AND LOCATIONS:
Overall Officials: David Furman, PhD, Principal Investigator — Chairman of the Scientific Advisory Board
Locations (2):
- United States (2):
  - La Follette Ob-Gyn & Aesthetics, Greenbrae, California
  - Herman Clinical Research, LLC, Suwanee, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veselkov K, Gonzalez G, Aljifri S, Galea D, Mirnezami R, Youssef J, Bronstein M, Laponogov I. HyperFoods: Machine intelligent mapping of cancer-beating molecules in foods. Sci Rep. 2019 Jul 3;9(1):9237. doi: 10.1038/s41598-019-45349-y. PMID 31270435
- [Background] Woo G, Fernandez M, Hsing M, Lack NA, Cavga AD, Cherkasov A. DeepCOP: deep learning-based approach to predict gene regulating effects of small molecules. Bioinformatics. 2020 Feb 1;36(3):813-818. doi: 10.1093/bioinformatics/btz645. PMID 31504186
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Damin AE, Nitrini R, Brucki SMD. Cognitive Change Questionnaire as a method for cognitive impairment screening. Dement Neuropsychol. 2015 Jul-Sep;9(3):237-244. doi: 10.1590/1980-57642015DN93000005. PMID 29213967
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Sayed N, Gao T, Ribshirani R, Hastie T, Cui L, Kuznetsova T, Rosenberg-Hasson Y, Ostan R, Monti D, Lehallier B, Shen-Orr S, Maecker HT, Dekker CL, Wyss-Coray T, Franceschi , Jojic V, Haddad F, Montoya JG, Wu JC and Furman D. An Inflammatory Clock Predicts Multi-morbidity, Immunosenescence and Cardiovascular Aging in Humans. (2019) bioRxiv 840363; doi: https://doi.org/10.1101/840363
- [Background] Bradley, C. L. A. R. E. The well-being questionnaire. Chur, Switzerland, Harwood Academic Publishers, 1994.
- [Background] Fung EB, Kwiatkowski JL, Huang JN, Gildengorin G, King JC, Vichinsky EP. Zinc supplementation improves bone density in patients with thalassemia: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2013 Oct;98(4):960-71. doi: 10.3945/ajcn.112.049221. Epub 2013 Aug 14. PMID 23945720
- [Background] Awad A, Zaglool AW, Ahmed SAA, Khalil SR. Transcriptomic profile change, immunological response and disease resistance of Oreochromis niloticus fed with conventional and Nano-Zinc oxide dietary supplements. Fish Shellfish Immunol. 2019 Oct;93:336-343. doi: 10.1016/j.fsi.2019.07.067. Epub 2019 Jul 25. PMID 31352117
- [Background] Guzman-Rivero M, Verduguez-Orellana A, Montano K, Cloetens L, Rojas E, Akesson B, Sejas E. The immune response in patients with cutaneous leishmaniasis and the influence of zinc supplementation. Biomed Pharmacother. 2015 Feb;69:56-62. doi: 10.1016/j.biopha.2014.11.006. Epub 2014 Nov 15. PMID 25661338
- [Background] Green JA, Lewin SR, Wightman F, Lee M, Ravindran TS, Paton NI. A randomised controlled trial of oral zinc on the immune response to tuberculosis in HIV-infected patients. Int J Tuberc Lung Dis. 2005 Dec;9(12):1378-84. PMID 16466061
- [Background] Guzman-Rivero, M., Verduguez-Orellana, A., Cordova, M., Maldonado, L., Medina, M., Sejas, E., & Åkesson, B. (2014). Effect of zinc on immune functions in patients with pulmonary tuberculosis. Biomedicine & Preventive Nutrition, 4(2), 245-250.
- [Background] Acevedo-Murillo JA, Garcia Leon ML, Firo-Reyes V, Santiago-Cordova JL, Gonzalez-Rodriguez AP, Wong-Chew RM. Zinc Supplementation Promotes a Th1 Response and Improves Clinical Symptoms in Fewer Hours in Children With Pneumonia Younger Than 5 Years Old. A Randomized Controlled Clinical Trial. Front Pediatr. 2019 Nov 14;7:431. doi: 10.3389/fped.2019.00431. eCollection 2019. PMID 31803694
- [Background] Ranasinghe P, Wathurapatha WS, Ishara MH, Jayawardana R, Galappatthy P, Katulanda P, Constantine GR. Effects of Zinc supplementation on serum lipids: a systematic review and meta-analysis. Nutr Metab (Lond). 2015 Aug 4;12:26. doi: 10.1186/s12986-015-0023-4. eCollection 2015. PMID 26244049
- [Background] Rosenkranz E, Hilgers RD, Uciechowski P, Petersen A, Plumakers B, Rink L. Zinc enhances the number of regulatory T cells in allergen-stimulated cells from atopic subjects. Eur J Nutr. 2017 Mar;56(2):557-567. doi: 10.1007/s00394-015-1100-1. Epub 2015 Nov 20. PMID 26589301
- [Background] Tsai YL, Ko WS, Hsiao JL, Pan HH, Chiou YL. Zinc sulfate improved the unbalanced T cell profiles in Der p-allergic asthma: An ex vivo study. Clin Respir J. 2018 Feb;12(2):563-571. doi: 10.1111/crj.12563. Epub 2016 Oct 23. PMID 27727525
- [Background] Salahuddin N, Ali F, Hasan Z, Rao N, Aqeel M, Mahmood F. Vitamin D accelerates clinical recovery from tuberculosis: results of the SUCCINCT Study [Supplementary Cholecalciferol in recovery from tuberculosis]. A randomized, placebo-controlled, clinical trial of vitamin D supplementation in patients with pulmonary tuberculosis'. BMC Infect Dis. 2013 Jan 19;13:22. doi: 10.1186/1471-2334-13-22. PMID 23331510
- [Background] Bischoff-Ferrari HA, Dawson-Hughes B, Stocklin E, Sidelnikov E, Willett WC, Edel JO, Stahelin HB, Wolfram S, Jetter A, Schwager J, Henschkowski J, von Eckardstein A, Egli A. Oral supplementation with 25(OH)D3 versus vitamin D3: effects on 25(OH)D levels, lower extremity function, blood pressure, and markers of innate immunity. J Bone Miner Res. 2012 Jan;27(1):160-9. doi: 10.1002/jbmr.551. PMID 22028071
- [Background] Rieder SA, Nagarkatti P, Nagarkatti M. Multiple anti-inflammatory pathways triggered by resveratrol lead to amelioration of staphylococcal enterotoxin B-induced lung injury. Br J Pharmacol. 2012 Nov;167(6):1244-58. doi: 10.1111/j.1476-5381.2012.02063.x. PMID 22646800
- [Background] Lu YJ, Jan YJ, Ko BS, Liang SM, Chen L, Wu CC, Chin CH, Kuo CC, Yet SF, Liou JY. Expression of Nik-related kinase in smooth muscle cells attenuates vascular inflammation and intimal hyperplasia. Aging (Albany NY). 2020 Apr 24;12(8):7511-7533. doi: 10.18632/aging.103104. Epub 2020 Apr 24. PMID 32330120
- [Background] Yang CJ, Lin CY, Hsieh TC, Olson SC, Wu JM. Control of eotaxin-1 expression and release by resveratrol and its metabolites in culture human pulmonary artery endothelial cells. Am J Cardiovasc Dis. 2011;1(1):16-30. Epub 2011 Apr 26. PMID 22254182
- [Background] Tan Y, Lim LH. trans-Resveratrol, an extract of red wine, inhibits human eosinophil activation and degranulation. Br J Pharmacol. 2008 Dec;155(7):995-1004. doi: 10.1038/bjp.2008.330. Epub 2008 Sep 8. PMID 18776917
- [Background] Singh NP, Hegde VL, Hofseth LJ, Nagarkatti M, Nagarkatti P. Resveratrol (trans-3,5,4'-trihydroxystilbene) ameliorates experimental allergic encephalomyelitis, primarily via induction of apoptosis in T cells involving activation of aryl hydrocarbon receptor and estrogen receptor. Mol Pharmacol. 2007 Dec;72(6):1508-21. doi: 10.1124/mol.107.038984. Epub 2007 Sep 14. PMID 17872969
- [Background] Mythri RB, Raghunath NR, Narwade SC, Pandareesh MDR, Sabitha KR, Aiyaz M, Chand B, Sule M, Ghosh K, Kumar S, Shankarappa B, Soundararajan S, Alladi PA, Purushottam M, Gayathri N, Deobagkar DD, Laxmi TR, Srinivas Bharath MM. Manganese- and 1-methyl-4-phenylpyridinium-induced neurotoxicity display differences in morphological, electrophysiological and genome-wide alterations: implications for idiopathic Parkinson's disease. J Neurochem. 2017 Nov;143(3):334-358. doi: 10.1111/jnc.14147. Epub 2017 Oct 3. PMID 28801915
- [Background] Roedel EQ, Cafasso DE, Lee KW, Pierce LM. Pulmonary toxicity after exposure to military-relevant heavy metal tungsten alloy particles. Toxicol Appl Pharmacol. 2012 Feb 15;259(1):74-86. doi: 10.1016/j.taap.2011.12.008. Epub 2011 Dec 16. PMID 22198552
- [Background] National Nutritional Foods Association, NNFA List of Dietary Supplement Ingredients In Use Before October 15, 1994 (April 26, 1996). Docket No.FDA-2005-P-0259 [Document ID: FDA-2005-P-0259-0012].
- [Background] Piotrowska H, Kucinska M, Murias M. Biological activity of piceatannol: leaving the shadow of resveratrol. Mutat Res. 2012 Jan-Mar;750(1):60-82. doi: 10.1016/j.mrrev.2011.11.001. PMID 22108298
- [Background] Fujioka N, Fritz V, Upadhyaya P, Kassie F, Hecht SS. Research on cruciferous vegetables, indole-3-carbinol, and cancer prevention: A tribute to Lee W. Wattenberg. Mol Nutr Food Res. 2016 Jun;60(6):1228-38. doi: 10.1002/mnfr.201500889. Epub 2016 May 23. PMID 26840393